CLINICAL TRIAL: NCT00811993
Title: Phase Ib Study To Evaluate The Safety Of Combining IGF-1R Antagonist R1507 With Multiple Standard Chemotherapy Drug Treatments In Patients With Advanced Malignancies
Brief Title: A Study of R1507 in Combination With Multiple Standard Chemotherapy Treatments in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO22068
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — RG-1507 monoclonal antibody; Bevacizumab; Capecitabine; Carboplatin; Cetuximab; Docetaxel; Erlotinib Hydrochloride; Etoposide; Gemcitabine; Irinotecan; Paclitaxel; Sorafenib; Temozolomide; Trastuzumab

ARMS (13):
- 1 (Experimental)
  Interventions: Drug: RG1507; Drug: erlotinib [Tarceva]; Drug: gemcitabine
- 10 (Experimental)
  Interventions: Drug: RG1507; Drug: temozolomide
- 11 (Experimental)
  Interventions: Drug: RG1507; Drug: bevacizumab [Avastin]; Drug: docetaxel
- 12 (Experimental)
  Interventions: Drug: RG1507; Drug: pemetrexel
- 13 (Experimental)
  Interventions: Drug: RO1507
- 2 (Experimental)
  Interventions: Drug: RG1507; Drug: bevacizumab [Avastin]; Drug: paclitaxel
- 3 (Experimental)
  Interventions: Drug: RG1507; Drug: carboplatin; Drug: etoposide
- 4 (Experimental)
  Interventions: Drug: RG1507; Drug: bevacizumab [Avastin]; Drug: mFOLFOX6
- 5 (Experimental)
  Interventions: Drug: RG1507; Drug: capecitabine [Xeloda]; Drug: trastuzumab [Herceptin]
- 6 (Experimental)
  Interventions: Drug: RG1507; Drug: sorafenib
- 7 (Experimental)
  Interventions: Drug: RG1507; Drug: bevacizumab [Avastin]; Drug: erlotinib [Tarceva]
- 8 (Experimental)
  Interventions: Drug: RG1507; Drug: cetuximab; Drug: irinotecan
- 9 (Experimental)
  Interventions: Drug: RG1507; Drug: bevacizumab [Avastin]; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: RG1507 — Starting dose of >=3mg/kg iv escalating to a maximum dose of <=16mg/kg iv, depending on dosing schedule in each combination treatment arm
  Arms: 1; 10; 11; 12; 2; 3; 4; 5; 6; 7; 8; 9
Drug: RO1507 — 27mg/kg iv, monotherapy
  Arms: 13
Drug: bevacizumab [Avastin] — as prescribed
  Arms: 11; 2; 4; 7; 9
Drug: capecitabine [Xeloda] — as prescribed
  Arms: 5
Drug: carboplatin — as prescribed
  Arms: 3; 9
Drug: cetuximab — as prescribed
  Arms: 8
Drug: docetaxel — as prescribed
  Arms: 11
Drug: erlotinib [Tarceva] — as prescribed
  Arms: 1; 7
Drug: etoposide — as prescribed
  Arms: 3
Drug: gemcitabine — as prescribed
  Arms: 1
Drug: irinotecan — as prescribed
  Arms: 8
Drug: mFOLFOX6 — as prescribed
  Arms: 4
Drug: paclitaxel — as prescribed
  Arms: 2; 9
Drug: pemetrexel — as prescribed
  Arms: 12
Drug: sorafenib — as prescribed
  Arms: 6
Drug: temozolomide — as prescribed
  Arms: 10
Drug: trastuzumab [Herceptin] — as prescribed
  Arms: 5

SUMMARY:
This study will evaluate the safety and tolerability of R1507 in combination with 12 distinct standard chemotherapy drug regimens and an additional R1507 monotherapy arm in patients with advanced malignant neoplasms.The 12 regimens will be tested in parallel. There are 3 subsets of patients who are eligible for the study: untreated, treated and requiring further treatment, or treated and failed and for whom adding R1507 represents a suitable treatment for their disease. All regimens will first test doses of R1507 which are less than the maximally administered dose, and if tolerated, the dose will be escalated in subsequent patients. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* malignant neoplasms;
* failed prior standard curative therapy;
* ECOG performance Status of 0 or 1;
* adequate bone marrow, hepatic and renal function;
* life expectancy greater than 8 weeks.

Exclusion Criteria:

* chemotherapy within 2 weeks of start of therapy;
* prior irradiation within 4 weeks prior to start of therapy;
* prior treatment with agents targeting IGF-IR inhibition, or other investigational agents;
* major surgery or significant traumatic injury within 2 weeks prior to study start;
* patients receiving concurrent antibody or immunotherapy;
* other exclusion criteria are related to specific treatment regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory parameters, vital signs | Throughout study

SECONDARY OUTCOMES:
Trough levels of R1507 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - Tucson, Arizona
  - San Francisco, California
  - Santa Monica, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Rochester, Minnesota
  - Chapel Hill, North Carolina
  - Houston, Texas